CLINICAL TRIAL: NCT04665336
Title: The Effect of Circadian Timing Program Created for Obese Individuals With Evening Chronotype on Obesity Management and Sleep Quality
Brief Title: The Effect of Circadian Timing Program on Obesity Management and Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Collaborators: Sakarya University (Other)
Responsible Party: Principal Investigator, Secil EKİZ ERİM, Research Assistant, Msc, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KOU
Record Dates: First submitted 2020-12-03; First posted 2020-12-11 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Obesity
Keywords: obese; chronotype; eveningness; circadian rhythm; sleep quality
MeSH Terms: conditions — Obesity; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group Lifestyle counseling (Experimental): Obese individuals with evening chronotype will be trained on sleep hygiene in order to create behavioral changes in line with circadian rhythms and an intervention program called "Circadian Timing Program" which was created by the researcher in line with the relevant literature will be implemented for 12 weeks. This program includes sleep hygiene recommendations and regulation of daylight exposure, sleep, meal, caffeine intake and exercise times. To determine participants' sleep times they will be asked to keep a sleep diary and sleep records will be taken with the smart bracelet. Participants will be given a password to access the research website. The website of the study will be used for the training, control, motivation and communication of the Participants.
  Interventions: Behavioral: Circadian Timing Program; Behavioral: Sleep Hygiene Training
- Control group (No Intervention): Participants will be asked to follow their normal daily lifestyle, maintain normal sleep and eating habits and no further instructions or suggestions will be provided during the study.

INTERVENTIONS:
Behavioral: Circadian Timing Program — Sleep hygiene training will be provided to the participants. They will be asked to make lifestyle changes according to the "Circadian Timing Program" created by the researcher.
  Arms: Intervention Group Lifestyle counseling
Behavioral: Sleep Hygiene Training — Sleep hygiene training will be given by the researcher. There will also be sleep hygiene training sections on the website.
  Arms: Intervention Group Lifestyle counseling

SUMMARY:
This study, it was aimed to examine the effect of circadian timing program created for obese individuals with evening chronotype on obesity management and sleep quality.

DETAILED DESCRIPTION:
The importance of chronotype, which reflects individual preferences in sleep timing and other behaviors, for obesity is mostly unknown. Morning types are more successful in long-term weight control than evening type chronotypes. Those with a sleep preference in the evening and a long sleep time have a higher rate of being overweight / obese than those with a morning preference and sufficient sleep time. Evening-type circadian preferences are indirectly related to food addiction. Individuals with the evening chronotype tend to have higher BMI and unhealthy eating habits.

Although a direct link between chronotype and obesity has not yet been demonstrated, based on the negative health consequences in evening chronotypes; In this study, it is assumed that success in obesity management will increase with well-timed circadian / sleep cycles, adequate sleep time and quality sleep in obese individuals with evening chronotype.

Therefore, in this study, it was aimed to examine the effect of circadian timing program created for obese individuals with evening chronotype on obesity management and sleep quality.

This study will be conducted in an experimental design, in a randomized controlled manner, in accordance with its purpose. The universe of the study will be obese individuals followed in Kocaeli University Hospital Obesity Outpatient Clinic. As a result of the power analysis performed to determine the sample size, the number of individuals in each group was determined as n = 18. The sample of the study will be 36 individuals in total. Participants will be selected to the intervention and control groups by simple randomization method.

ELIGIBILITY:
Inclusion Criteria:

* Being followed in Kocaeli University Hospital Obesity Outpatient Clinic
* Being an obese adult (BMI ≥ 30.0 kg / m²)
* Being in the age group of 18 and over
* Having the evening chronotype (Individuals with a late sleep period)
* Having a calorie-based diet according to body mass index and adapting to his diet
* To know how to read and write
* Not to have sensory losses such as sight and hearing
* Not being physically, cognitively or mentally obstructed to participate in the research
* To be open to communication and cooperation
* To have and use internet access
* Having a smart phone

Exclusion Criteria:

* Insomnia, regular sleep, shift work
* Traveling in time zones in the last 4 weeks
* Having an eating or psychiatric disorder
* Alcohol addiction
* Nursing mothers who are pregnant or lactating (giving birth in the past two years)
* Do not use antiobesity medication
* New diagnosis of hyperlipidemia and diabetes and drug initiation (in dose adjustment for less than 3 months)
* Heavy exercise or a sedentary lifestyle
* Being on insulin therapy
* Having a risk of hypoglycemia
* Having Chronic Obstructive Pulmonary Disease, Sleep Apnea, Celiac, Severe Anemia, disease / illnesses

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) from Baseline at 12 Week | Change between day 1 and week 12 of the study.
  Measurements will be made with body analysis device and height meter in the outpatient clinic. The Body-Mass Index is calculated by dividing the person's weight in kilograms by the square of the person's height in meters (kg / m²). Change = (Week 12 Measurement- Baseline Measurement).
Change in waist and hip circumference from Baseline at 12 Week | Change between day 1 and week 12 of the study.
  Waist and hip circumference is measured with a tape measure, graduated in centimetres, . The waist-hip ratio is calculated as waist measurement divided by hip measurement W ÷ H. Change = (Week 12 Measurement- Baseline Measurement).
Change from Baseline in Sleep Quality on The Pittsburgh Sleep Quality Index (PUKI) at Week 12. | Baseline and Week 12
  PUKI is a scale that can define the quality of sleep as "good or bad". Change = (Week 12 Measurement- Baseline Measurement).

SECONDARY OUTCOMES:
Change in Quality of Life from Baseline at 12 Week. | Baseline and Week 12
  In the Impact of Weight on Quality of Life Instrument (IWQOL-Lite)
Change in Sleepiness from Baseline at 12 Week. | Baseline and Week 12
  In the Epworth Sleepiness Scale (ESS) the lowest score that can be obtained from the scale

CONTACTS AND LOCATIONS:
Overall Officials: Havva Sert, Assoc. Prof., Study Director — Sakarya University
Locations (1):
- Kocaeli University, İzmit, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kolotkin RL, Crosby RD, Kosloski KD, Williams GR. Development of a brief measure to assess quality of life in obesity. Obes Res. 2001 Feb;9(2):102-11. doi: 10.1038/oby.2001.13. PMID 11316344
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Izci B, Ardic S, Firat H, Sahin A, Altinors M, Karacan I. Reliability and validity studies of the Turkish version of the Epworth Sleepiness Scale. Sleep Breath. 2008 May;12(2):161-8. doi: 10.1007/s11325-007-0145-7. PMID 17922157
- [Background] Horne JA, Ostberg O. A self-assessment questionnaire to determine morningness-eveningness in human circadian rhythms. Int J Chronobiol. 1976;4(2):97-110. PMID 1027738
- [Background] Ross KM, Graham Thomas J, Wing RR. Successful weight loss maintenance associated with morning chronotype and better sleep quality. J Behav Med. 2016 Jun;39(3):465-71. doi: 10.1007/s10865-015-9704-8. Epub 2015 Dec 10. PMID 26660638
- [Background] Nohara K, Yoo SH, Chen ZJ. Manipulating the circadian and sleep cycles to protect against metabolic disease. Front Endocrinol (Lausanne). 2015 Mar 23;6:35. doi: 10.3389/fendo.2015.00035. eCollection 2015. PMID 25852644
- [Derived] Ekiz Erim S, Sert H. The effect of circadian timing program for evening-chronotype individuals with obesity on obesity management and sleep quality: A randomized controlled trial. Sleep Med. 2024 Jul;119:58-72. doi: 10.1016/j.sleep.2024.04.017. Epub 2024 Apr 16. PMID 38652930